CLINICAL TRIAL: NCT07225985
Title: Salvage Treatment With Bendamustine and Pralatrexate Followed Immediately by Reduced-Intensity Conditioning (RIC) Allogeneic Hematopoietic Cell Transplantation (Prala-Benda/RIC) for Adults With T Cell Lymphomas: A Phase 1/2 Study
Brief Title: Pralatrexate With Bendamustine and Total-Body Irradiation Followed by Donor Stem Cell Transplant for the Treatment of Relapsed or Refractory T-Cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125830; NCI-2025-07661 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Bendamustine Hydrochloride; 10-propargyl-10-deazaaminopterin; Biopsy; X-Rays; Spinal Puncture; Magnetic Resonance Spectroscopy; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pralatrexate, bendamustine, TBI, PBSC HCT) (Experimental): Patients receive pralatrexate IV over 3-5 minutes on day -6, bendamustine IV over 60 minutes on days -5, -4, and -3, and TBI on day -1 or 0. Patients then undergo PBSC HCT on day 0. Patients also undergo ECHO or MUGA and lumbar puncture during screening, PET-CT, MRI, bone marrow biopsy/aspiration, and blood sample collection throughout the study. In addition, patients may undergo chest X-rays as clinically indicated.
  Interventions: Drug: Bendamustine; Drug: Pralatrexate; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Total-Body Irradiation; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Bendamustine — Given IV
  Other Names: SDX 105; SDX-105; SDX105
Drug: Pralatrexate — Given IV
  Other Names: 10-propargyl-10-deazaaminopterin; Difolta; Folotyn; PDX
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy/aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy/aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Chest Radiography — Undergo chest X-rays
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC HCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I/II trial studies the side effects and best dose of pralatrexate in combination with bendamustine and total-body irradiation (TBI) followed by a donor stem cell transplant in treating patients with T-cell non-Hodgkin lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Pralatrexate may block the growth of cancer cells and cause them to die. It is a type of dihydrofolate reductase (DHFR) inhibitor. Bendamustine may damage the DNA in cancer cells and cause them to die. It is a type of alkylating agent and a type of antimetabolite. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. TBI is a type of radiation therapy that is given to the entire body. Giving pralatrexate with bendamustine and TBI before a donor stem cell transplant may help kill cancer cells in the body and help make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow.

DETAILED DESCRIPTION:
OUTLINE:

This is a phase I dose-escalation study of pralatrexate in combination with bendamustine and TBI followed by a phase II expansion study.

Patients receive pralatrexate intravenously (IV) over 3-5 minutes on day -6, bendamustine IV over 60 minutes on days -5, -4, and -3, and TBI on day -1 or 0. Patients then undergo peripheral blood stem cell (PBSC) HCT on day 0. Patients also undergo echocardiography (ECHO) or multi-gated acquisition scan (MUGA) and lumbar puncture during screening, positron emission tomography-computed tomography (PET-CT), magnetic resonance imaging (MRI), bone marrow biopsy/aspiration, and blood sample collection throughout the study. In addition, patients may undergo chest X-rays as clinically indicated.

After completion of study treatment, patients are followed up at 6 months, at 1 year, and at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with an HCT-Comorbidity Index (CI) ≤ 5 for patients over 60 years
* T-cell non-Hodgkin lymphoma (T-NHL) (2022 World Health Organization [WHO] criteria) including primary cutaneous T-NHL that is in untreated or unsuccessfully treated first or subsequent relapse. Patients in morphologic remission (i.e. < 5% blasts in the bone marrow, if involved) but evidence of minimal residual disease (MRD) by positron emission tomography-computed tomography (PET-CT), multiparameter flow cytometry, cytogenetics/fluorescence in situ hybridization (FISH), or molecular means will be eligible for trial participation
* The use of bridging chemotherapy prior to initiation of study treatment is allowed. Patients with symptoms/signs of hyperleukocytosis, white blood cells (WBC) > 100,000/µL, or with concern for other complications of high tumor burden of high tumor dynamics (e.g. disseminated intravascular coagulation) can be treated with leukapheresis or may receive a cycle of salvage chemotherapy prior to start of study treatment
* Karnofsky score ≥ 70; Eastern Cooperative Oncology Group (ECOG) 0-1
* Adequate cardiac function defined as absence of decompensated congestive heart failure and/or uncontrolled arrhythmia and left ventricular ejection fraction ≥ 45%
* Bilirubin ≤ 2.5 x institutional upper limit of normal unless elevation is thought to be due to hepatic infiltration by acute myeloid leukemia (AML), Gilbert's syndrome, or hemolysis
* Adequate pulmonary function defined as absence of oxygen (O2) requirements and either diffusion capacity of the lung for carbon monoxide (DLCO) corrected ≥ 70%mmHg or DLCO corrected 60-69%mmHg and partial pressure of oxygen (pO2) ≥ 70mmHg
* Creatinine clearance ≥ 60 mL/min
* Prior autologous HCT is permissible if relapse occurred > 6 months after HCT
* A human leukocyte antigen (HLA)-matched sibling/unrelated donor mismatched unrelated donor or haploidentical donor for collection of stimulated peripheral blood stem cells must be identified and readily available
* If the patient has received pralatrexate or bendamustine before and has been sensitive to this regimen, defined as MRD negative complete response (CR) immediately after receiving the treatment and which lasts ≥ 1 year, eligibility will be determined on a case-by-case basis by the study principal investigator (PI)
* Ability to understand and sign a written informed consent document (or legal representative)
* RELATED DONOR: Related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1. Phenotypic identity must be confirmed by high-resolution typing
* MATCHED UNRELATED DONOR: Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR
* MATCHED UNRELATED DONOR: Mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
* MATCHED UNRELATED DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment. The recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT. If the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained. The donor should be excluded if any of the cytotoxic cross match assays are positive. For those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results. A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion.
* MATCHED UNRELATED DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed.
* MISMATCHED UNRELATED DONOR: HLA-matching must be based on results of high resolution typing at HLA-A, -B, -C, -DRB1, and -DQ
* MISMATCHED UNRELATED DONOR: Mismatch for one HLA class I antigen with or without an additional mismatch for one HLA-class I allele but matched for HLA-DRB1 and HLA-DQ
* MISMATCHED UNRELATED DONOR: Mismatched for two HLA class I alleles but matched for HLA-DRB1 and HLA-DQ
* MISMATCHED UNRELATED DONOR: HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen/allele mismatch
* MISMATCHED UNRELATED DONOR: If the patient is homozygous at the mismatch HLA class I locus or II locus, the donor must be heterozygous at that locus and one allele must match the patient (i.e., patient is homozygous A*01:01 and donor is heterozygous A*01:01, A*02:01). This mismatch will be considered a one-antigen mismatch for rejection only
* HAPLOIDENTICAL DONOR: Donors must be haploidentical relatives of the patients. Donor-recipient compatibility will be tested through HLA typing at high resolution for the HLA loci (-A, -B, -C, -DRB1, -DQB1). Donor and recipient should share at least 5/10 HLA loci
* HAPLOIDENTICAL DONOR: Age ≥ 18 years
* HAPLOIDENTICAL DONOR: Weight ≥ 40 kg
* HAPLOIDENTICAL DONOR: Donor must meet the selection criteria as defined by the Foundation of the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines
* HAPLOIDENTICAL DONOR: In case of more available haploidentical donors, selection criteria should include, in this order:

  * For cytomegalovirus (CMV) seronegative recipients, a CMV seronegative donor
  * Red blood cell compatibility

    * Red blood cell (RBC) cross match compatible
    * Minor ABO incompatibility
    * Major ABO incompatibility

Exclusion Criteria:

* Active central nervous system (CNS) disease
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with antimicrobials and/or controlled or stable. Patients with fever thought to be likely secondary to myeloid malignancy are eligible
* Known hypersensitivity or contraindication to any study drug used in this trial
* Pregnancy or lactation
* Concurrent treatment with any other approved or investigational anti-lymphoma agent at the time of starting conditioning
* HAPLOIDENTICAL DONOR: Since detection of anti-donor-specific antibodies (anti-DSA) is associated with higher graft rejection rate, patients will be screened for anti-DSA pre-transplant. Patient with DSA mean fluorescent intensity (MFI) < 5000 after desensitization treatment, will be considered eligible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events and treatment emergent serious adverse events | From pralatrexate dosing on day -6 to 100 days post-transplant
  In addition, clinically significant laboratory abnormalities, changes in vital signs, and changes in physical examination following allogeneic hematopoietic cell transplantation (allo-HCT).

SECONDARY OUTCOMES:
Proportion of enrolled patients with T-cell non-Hodgkin lymphoma who successfully proceed to allo-HCT | Up to 2 years post-transplant
  Will compare it with the historical rate of 31%. An exact one-sample (one-sided) binomial test will be used, with a nominal significance level of α = 0.15.
Cumulative incidence of graft-versus-host disease (GVHD) | Up to 1 year post-transplant
  Group comparisons will be performed using Gray's test, and multivariable analyses will be conducted using cause-specific Cox model to assess the effect of covariates. The cumulative incidence of acute GVHD (grades II-IV and III-IV) by day +100 and chronic GVHD at 1 year will be estimated using the cumulative incidence function.
Incidence of grade II-IV acute GVHD | Up to day 100 post-transplant
  Group comparisons will be performed using Gray's test, and multivariable analyses will be conducted using cause-specific Cox model to assess the effect of covariates.
Incidence of chronic GVHD requiring systemic immunosuppressive therapy | At 1 year post-transplant
  Group comparisons will be performed using Gray's test, and multivariable analyses will be conducted using cause-specific Cox model to assess the effect of covariates.
Disease response rate | At day 100 post-transplant
  Proportion and counts will be calculated with an exact 95% confidence intervals.
Duration of remission from response until documented relapse or progression | From response until documented relapse or progression, per disease-specific response criteria up to 2 years post-transplant
Proportion of donor chimerism ≥ 90% in peripheral blood CD3+ and CD33+ cell lines | Up to day 80 post-transplant
  Proportion and counts will be calculated with an exact 95% confidence intervals. Donor chimerism will be summarized by the observed levels and levels categorized as ≥ 95%, 50% - 94%, 5% - 49%, or < 5%.
Disease-free survival | From day 0 (date of graft infusion) to the first of: Relapse/progression of the underlying disease, or death from any cause, assessed up to 1 year post-transplant
  Defined as the proportion of patients who are alive and free of disease relapse/progression at 1 year (365 days) after day 0. Proportion and counts will be calculated with an exact 95% confidence intervals. Kaplan-Meier method will be used to estimate the median with 95% confidence intervals. Log-rank test will be used for group comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Iovino, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No